CLINICAL TRIAL: NCT00667667
Title: Effect of Whole Body Vibration Training on Two Different Devices on Osteoporotic Risk Factors in Postmenopausal Women. A Randomized Controlled Trial.
Brief Title: Effects of Whole Body Vibration on Postmenopausal Risk-factors in Elderly Women
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Elsbeth-Bonhoff-Stiftung, Berlin (Unknown)
Responsible Party: Principal Investigator, Wolfgang Kemmler, Principal Investigator, University of Erlangen-Nürnberg Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OFZ-Elvis-II
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Postmenopausal
Keywords: whole body vibration; exercise; postmenopausal; BMD; bone; elderly females; Caucasian race
MeSH Terms: conditions — Motor Activity | interventions — Health; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): vertical vibration device (using Vibrafit whole body vibration platforms)
  Interventions: Device: vertical vibration device (Vibrafit whole body vibration platform)
- 2 (Active Comparator): side-alternating vibration device (using Board 3000 whole body vibration platforms)
  Interventions: Device: side alternating vibration device (Board 3000 whole body vibration platform)
- 3 (Sham Comparator): wellness-control group
  Interventions: Behavioral: stretching and wellness (control group)

INTERVENTIONS:
Device: vertical vibration device (Vibrafit whole body vibration platform) — 3 sessions/week 15 min each, leg exercises performed on whole body vibration platforms with vertical device
  Arms: 1
Device: side alternating vibration device (Board 3000 whole body vibration platform) — 3 sessions/week 15 min each, leg exercises performed on whole body vibration platforms with side alternating device
  Arms: 2
Behavioral: stretching and wellness (control group) — 2x10 weeks with 1 session/week of low volume, low intensity wellness training over 12 months
  Arms: 3

SUMMARY:
There is general agreement that physical exercise can positively influence osteoporotic fracture risk along two pathways: first by reducing the risk of falls via an improvement of fall related neuromuscular abilities; second by increasing bone strength.

Whole body vibration (WBV) training has recently been proposed as a new approach for prevention and treatment of osteoporosis. Animal studies have shown evidence that WBV may be an effective method to improve bone mass, architecture and strength. However, the results of human WBV training studies are rather heterogeneous.

In the Erlangen Longitudinal Vibration Study II (ELVIS II), a randomized, controlled 12 month lasting study the investigators determine the effect of a thrice weekly WBV training on two different devices on the osteoporotic risk factors: bone mineral density, falls and neuromuscular performance. Particular the investigators compare a bipedal vertical oscillating Plate with a plate which rotates around a central axis leading to a side-alternating loaning.

ELIGIBILITY:
Inclusion Criteria:

* females 60 - 75 years old
* caucasian race

Exclusion Criteria:

* CHD-diseases
* thrombosis, embolism
* fractures at lumbar spine or hip
* secondary osteoporosis
* hyperparathyroidism
* medication, diseases with impact on muscle or bone
* hip or knee implant

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2008-04; Primary Completion 2009-06 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density | Baseline, 12 months

SECONDARY OUTCOMES:
muscle strength | baseline, 12 months
Quality of life | baseline, 12 month
falls | daily over 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Simon O von Stengel, PhD, Principal Investigator — University of Erlangen-Nürnberg Medical School; Wolfgang K Kemmler, PhD, Study Chair — Instiute of Medical Physics; Willi A Kalender, Prof., PhD, Study Director — University of Erlangen-Nürnberg Medical School
Locations (1):
- Institute of Medical Physics, University of Erlangen-Nurnberg, Erlangen, Germany

REFERENCES:
- [Background] von Stengel S, Kemmler W, Kalender WA, Engelke K, Lauber D. Differential effects of strength versus power training on bone mineral density in postmenopausal women: a 2-year longitudinal study. Br J Sports Med. 2007 Oct;41(10):649-55; discussion 655. doi: 10.1136/bjsm.2006.033480. Epub 2007 Jun 5. PMID 17550916
- [Background] Stengel SV, Kemmler W, Pintag R, Beeskow C, Weineck J, Lauber D, Kalender WA, Engelke K. Power training is more effective than strength training for maintaining bone mineral density in postmenopausal women. J Appl Physiol (1985). 2005 Jul;99(1):181-8. doi: 10.1152/japplphysiol.01260.2004. Epub 2005 Mar 3. PMID 15746294
- [Background] Kemmler W, Lauber D, Weineck J, Hensen J, Kalender W, Engelke K. Benefits of 2 years of intense exercise on bone density, physical fitness, and blood lipids in early postmenopausal osteopenic women: results of the Erlangen Fitness Osteoporosis Prevention Study (EFOPS). Arch Intern Med. 2004 May 24;164(10):1084-91. doi: 10.1001/archinte.164.10.1084. PMID 15159265
- See also: homepage of the Institute of Medical Physics — http://www.imp.uni-erlangen.de/